CLINICAL TRIAL: NCT04413630
Title: Therapeutic Effects of Family-centered Workshops for Toddlers With Speech and Language Developmental Delay
Brief Title: Workshops for Toddlers With Speech and Language Developmental Delay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SKH-109
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Developmental Delay
Keywords: family workshop
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Intervention Model Description: Intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): family workshop
  Interventions: Other: family workshop

INTERVENTIONS:
Other: family workshop — The family workshop with 5 courses, with 6 families in one course The intervention of one course; 2 hours per session, one time per week, for a total of 6 weeks

SUMMARY:
The purpose of this study is to identify the therapeutic effects of family workshops on speech and language developmentally delayed children and their family

DETAILED DESCRIPTION:
The family workshop with 5 courses, 6 families in one course, a 2-hour session per week, for 6 weeks.

Effects:

1. Investigate the therapeutic effects of the workshop for the toddlers with developmental delay
2. Investigate the therapeutic effects of the workshop for the parents of toddlers with developmental delay

ELIGIBILITY:
Inclusion Criteria:

* 18 to 36 months old children with speech and language developmental delay with or without delay in gross motor, fine motor, cognition, and emotional or social function

the availability of toddlers and their parents to attend one 2-hour session of the workshop per week for 6 weeks

Exclusion Criteria:

* Less than 18 months old or older than 36 months old

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 122 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Chinese Communicative Developmental Inventory | scores change from baseline to 6 weeks after treatment, higher scores mean a better outcome
  assess communication and language function of children

SECONDARY OUTCOMES:
Peabody Developmental Motor Scales | scores change from baseline to 6 weeks after treatment, higher scores mean a better outcome
  assess fine motor function of children
Pediatric Outcomes Data Collection Instrument | scores change from baseline to 6 weeks after treatment, higher scores mean a better outcome
  measure the functional performance of children
Child Health Questionnaire-Parent Form 28 | scores change from baseline to 6 weeks after treatment, higher scores mean a better outcome
  assess the health status of children
Pediatric Quality of Life Inventory-Geriatric Core Scales | scores change from baseline to 6 weeks after treatment, higher scores mean a better outcome
  measure the quality of life of children
Caregiver Strain Index | scores change from baseline to 6 weeks after treatment, higher scores mean a worse outcome
  assess family strain
Impact on Family Scale | scores change from baseline to 6 weeks after treatment, higher scores mean a worse outcome
  assess the effects of a child's illness of the function of the family system
Pediatric Quality of Life Inventory-Family Impact Module | scores change from baseline to 6 weeks after treatment, higher scores mean a better outcome
  assess the impact of pediatric conditions on family function and quality of life
World Health Organization Quality of Life Brief Version | scores change from baseline to 6 weeks after treatment, higher scores mean a better outcome
  evaluate parents' quality of life
Parental satisfaction questionnaire | after completion of 6 weeks of workshop
  assess the parents' subjective satisfaction to the whole workshop itself, score ranges from 0 to 100, higher scores mean a higher satisfaction
Emotional Competency Rating Scales | scores change from baseline to 6 weeks after treatment
  assess emotional function of children, higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No